CLINICAL TRIAL: NCT00511693
Title: Regional Osteoporosis Coordinator Knowledge Exchange Trial
Brief Title: Osteoporosis Coordinator for Low Volume Community Hospitals
Acronym: ROCKET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ontario Ministry of Health and Long Term Care (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: TRI REB 07-029
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2007-08-07 (Estimated); Status verified 2007-07

CONDITIONS: Osteoporosis; Fragility Fractures
Keywords: fragility fracture; management of osteoporosis; osteoporosis coordinator; small volume hospitals
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): hospitals randomly allocated to receive physician and patient osteoporosis recommendations from the regional coordinator
  Interventions: Behavioral: centralized osteoporosis coordinator
- 2 (Active Comparator): hospitals randomly allocated to receive falls prevention advice
  Interventions: Behavioral: fall prevention

INTERVENTIONS:
Behavioral: centralized osteoporosis coordinator — The regional osteoporosis coordinator will phone fracture patients and counsel them about their risk of osteoporosis, reiterating messages in the print material. The coordinator will also follow-up with family physicians by phone and send them a patient-specific reminder that informs them that their patient has experienced a fracture and they are at high risk for future fracture. As part of the reminder, a set of evidence-based recommendations about appropriate BMD testing and treatment based on the recent Canadian guidelines will be included. If the patient does not have a family physician, the regional osteoporosis coordinator will facilitate referral to the MOP.
  Arms: 1
Behavioral: fall prevention — Fracture patients from hospitals receiving falls prevention advice will also be called by the osteoporosis regional coordinator. The patient will receive educational material and telephone counseling regarding fall prevention. During the call, patients will be encouraged to visit their family physician for fracture follow-up. They will not receive counseling or educational materials about osteoporosis at this time. Patients in the falls prevention group will receive the physician and patient osteoporosis program six months post-fracture.
  Arms: 2

SUMMARY:
A Regional Osteoporosis Coordinator located at Women's College Hospital will follow-up with low trauma fracture patients from 30 smaller community hospitals across Ontario. To evaluate whether this quality improvement program can increase post-fracture osteoporosis care in these individuals, hospitals will be randomized to receive osteoporosis specific recommendations or falls prevention advice. Patients will be asked to complete two short telephone surveys about their recent fracture, risk factors, osteoporosis knowledge and diagnostic and treatment history. All patients in the falls prevention advice group will receive the osteoporosis specific recommendations 6 months after their fracture.

DETAILED DESCRIPTION:
A. Background and Rationale. Despite the availability of proven safe and effective treatment options, the majority of patients with low trauma fracture are under-investigated and under-treated, indicating that treatment for osteoporosis after fracture is less than optimal. Most of the published studies on interventions using a coordinator recruited patients from one or a few academic centres or health maintenance organization. However, in Ontario, one-third of fracture patients are treated in non-academic centres and hospitals which have no dedicated osteoporosis fracture clinic coordinator and are underserviced for osteoporosis specialists. It remains unclear whether the impact will be as great for smaller centres where the coordinator function is centralized across multiple centres; hence the need for this trial.

B. Objectives 1. The primary objective is to evaluate if a quality improvement program including physician and patient osteoporosis recommendations from a regional osteoporosis coordinator will increase the proportion of individuals with a low trauma fracture who receive appropriate management for osteoporosis compared to those who receive only falls prevention advice.

2. A secondary objective is to determine if the above program will result in changes in perceived susceptibility, osteoporosis knowledge and use of supplements compared to those who receive only falls prevention advice.

C. Methods. Design: cluster randomized controlled trial (hospitals=cluster site) with the outcome assessors and data analyst blinded to group allocation.

Patient population: patients 40 years old and over (men and women) presenting with a low trauma fracture of the hip, forearm/wrist, rib(s), sternum, thoracic and lumbar spine, shoulder, upper arm, pelvis, lower leg and ankle. Hospitals that treat more than 40 patients/year and have no dedicated fracture clinic coordinator in their Emergency Department/Fracture Clinic will be considered.

Hospital recruitment: out of 63 hospitals 30 will be recruited (15 as intervention and 15 control); 20 patients from each hospital will be identified with the expectation that 10 will consent to the study, for a total sample size of 300 patients.

Intervention: provide evidenced-based recommendations and having a centralized osteoporosis coordinator follow-up with fracture patients and their physicians to provide information about fracture risk and osteoporosis treatment as part of educational outreach, assist with ordering BMD test and arranging consultation to Multidisciplinary Osteoporosis Program (MOP) via telehealth if required. For the control sites the same process will be followed for identifying fracture patients. They will receive educational material and telephone counseling regarding fall prevention and home safety and will be encouraged to visit their family physician.

Data collection. Patients will be identified from NACRS database. Baseline data will be collected by the osteoporosis coordinator. The questionnaire will be similar to "Fracture Clinic OP Screening Program". Follow-up data will be collected by a research assistant who will call consenting patients.

Data Analysis. The analysis of primary and secondary outcome measures will compare the intervention and control groups and will be carried out at the level of the cluster (hospital), based on the standard two-sample t-test with 2(k-1) degrees of freedom, where k is the number of sites in each group (α= 0.05, power=1-β).

D. Future implications. This trial will increase our understanding of how to implement care delivery models in communities in terms of resources, services and patient and provider preferences. At the health system level this trial will have direct relevance to Ontario's Osteoporosis Strategy. The findings will be used by decision-makers to determine if hospitals with no dedicated osteoporosis coordinator should be provided access to a centralized fracture coordinator. At the provider and patient level the trial will increase access to osteoporosis care and treatment utilization, along with awareness and knowledge regarding osteoporosis treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Cluster site (hospital) level: Hospitals with no dedicated osteoporosis coordinator that treat more than 60 patients/year in their Emergency Department and who have a Telehealth studio.
2. Patient level: Patients 40 years old and over (men and women) presenting with a low trauma fracture of the hip, forearm and wrist, rib(s), sternum, thoracic and lumbar spine, shoulder and upper arm, pelvis, lower leg and ankle. Subjects without previous medication as well as subjects on osteoporosis medication and presenting with a fracture will be included.

Exclusion Criteria:

1. Hospitals that have an Osteoporosis Strategy fracture clinic coordinator
2. Fractures associated with major trauma; fractures due to malignancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-06; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
proportion of patients from the intervention group as compared to the control group that had "appropriate management" based on a composite of undergoing a BMD test and starting therapy within 6 months of fracture. | 1.5 years

SECONDARY OUTCOMES:
osteoporosis knowledge, perceived susceptibility, self-efficacy, preventive behaviors | 1.5 years
participants' experience and perceptions of future fracture risk; their understanding of the educational materials and acceptance of recommended treatment plans. | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan B Jaglal PhD, Principal Investigator — Toronto Rehabilitation Institute, University of Toronto; Oana S Donescu MD PhD, Study Director — Toronto Rehabilitation Institute, University of Toronto
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jaglal SB, Donescu OS, Bansod V, Laprade J, Thorpe K, Hawker G, Majumdar SR, Meadows L, Cadarette SM, Papaioannou A, Kloseck M, Beaton D, Bogoch E, Zwarenstein M. Impact of a centralized osteoporosis coordinator on post-fracture osteoporosis management: a cluster randomized trial. Osteoporos Int. 2012 Jan;23(1):87-95. doi: 10.1007/s00198-011-1726-7. Epub 2011 Jul 16. PMID 21779817